CLINICAL TRIAL: NCT01416467
Title: Characterization of the Patient Population With Galactosialidosis
Acronym: CPPGAL
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Assisi Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPPGAL; R01DK095169 (NIH)
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Galactosialidosis
Keywords: lysosomal storage disease; AAV vector; gene transfer; disease characterization
MeSH Terms: conditions — Neuraminidase deficiency with beta-galactosidase deficiency; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood for PPCA gene mutation and AAV2 and AAV8 antibody titer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The late infantile form of galactosialidosis is potentially amenable to treatment by gene transfer with an adeno-associated viral vector encoding Protective Protein Cathepsin A (PPCA) or by infusion of purified protein. The published literature contains limited descriptions of the disease nor is it known how many patients with the disorder are potentially available for protocol enrollment. This preliminary study is designed to define the demographics and clinical characteristics of the patient population with galactosialidosis. Individuals for whom DNA diagnosis has been performed at St. Jude Children's Research Hospital (SJCRH) will be contacted telephonically to learn their current status. In addition, a letter requesting information regarding patients with galactosialidosis will be sent to all pediatric geneticists throughout the United States. Selected physicians with expertise in lysosomal storage diseases throughout the world will also be contacted. Foundations and Associations for the lysosomal storage disorders will also be contacted in an effort to identify additional potential patients with galactosialidosis. The information to be collected in this preliminary study will facilitate development of specific eligibility criteria for future therapeutic studies.

DETAILED DESCRIPTION:
Individual patient/families will be interviewed by telephone to learn basic demographic information and disease status. Medical records will be requested from primary care providers to provide further information regarding their disorder. Individual patients identified through our survey of pediatric geneticists or via the disease foundations or associations will be sent a letter describing our purpose and which includes a consent form for a subsequent telephonic interview. Their medical records will also be requested.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with suspected or confirmed molecular diagnosis of galactosialidosis who are ≥ 6 months of age.

Exclusion Criteria:

* Individuals with a lysosomal storage disorder who have been shown to have a mutation in a gene other than that encoding PPCA.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with suspected or diagnosed galactosialidosis.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-02-08 (Actual); Primary Completion 2012-04-12 (Actual); Study Completion 2012-04-12 (Actual)

PRIMARY OUTCOMES:
Mean, median and standard deviation of age distribution of patients with galactosialidosis. | At enrollment
  The clinical and demographic data will be tabulated and analyzed for age distribution and disease manifestations with a goal of defining eligibility criteria for future therapeutic protocols.

SECONDARY OUTCOMES:
Number and type of PPCA gene mutations in patients with galactosialidosis. | At enrollment
  The genotyping data will be tabulated and analyzed to determine the spectrum of mutations that result in the late infantile form of galactosialidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Reiss, MD, Principal Investigator — St. Jude Children's Research Hospital; Alessandra D'Azzo-Grosveld, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols